CLINICAL TRIAL: NCT05933369
Title: The Impact of Clinical Pharmacist Intervention on Asthmatic Patient's Outcomes at the University of Gondar Comprehensive and Specialized Hospital, Northwest Ethiopia, 2022: A Randomized Controlled Trial
Brief Title: The Impact of Clinical Pharmacist Intervention on Asthmatic Patient's Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Gondar (Other)
Responsible Party: Principal Investigator, Eden Abetu Mehari, Principal investigator, University of Gondar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASTHMA-PHAR
Record Dates: First submitted 2023-03-21; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Asthma
Keywords: ASTHMA-PHAR; Asthma; Clinical pharmacist led intervention
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor assessing patient outcomes will be blind. The participants and the intervention providers (Clinical pharmacists) will not be blind for patient assignment to one of the trial groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients in the intervention group will receive a protocol-defined clinical pharmacist intervention at the start of the study and at the 1- , 3 and 6-month follow-up visits.
  Interventions: Behavioral: Clincal pharmacist intervention
- Control (No Intervention): Patients in the control group will receive the usual pharmacist care.

INTERVENTIONS:
Behavioral: Clincal pharmacist intervention — Patients in the intervention group will receive a protocol-defined intervention at the start of the study and at the 1- , 3 and 6-month follow-up visits for education on disease and treatment 40 minutes, administration and dosage 6 minutes, drug interaction and other drug therapy problems 20 minutes for a total of 66 minutes. The intervention will include education about asthma triggers and the need of minimizing them, asthma symptoms, warning signs, proper inhalation use technique, cigarette smoking cession when appropriate, the need of adherence and they will also counseled to wash their mouth after the use of controller medications. In addition, pharmaceutical care evaluation will be carried out and any drug therapy problems will be addressed accordingly and finally every intervention provided will be recorded.
  Arms: Intervention

SUMMARY:
The goal of this trial is to determine whether or not clinical pharmacist led intervention for 3 months improves asthma control of asthmatic patients' outcomes as compared to the usual care 2023. The main question it aims to answer is does clinical pharmacist led interventions improve patient outcomes of asthmatic patients? Patients in the intervention group will receive a protocol-defined intervention at the start of the study and at the 1- , 3 and 6-month follow-up visits. Patients in the control group will receive the usual pharmacist care.

DETAILED DESCRIPTION:
There are poor patient outcomes in the study area as it is evident in previous studies where almost ninety five percent of patients had not well controlled Asthma. Moreover, the rate of non-adherence to inhalational anti asthmatics is high and more than half of asthmatic patients received inappropriate treatment. All those poor patient outcomes can be easily prevented and those studies have recommended that patient education and proper patient consultation to optimize the benefits of treatment by integrating clinical pharmacists. Thus, pharmacists are at sealing point at which most of medication information must be provided if a conducive system is created which can greatly improve patient's treatment outcome.

This study will generate strong evidence on the impact of clinical pharmacists at improving asthma control. It will also be an excellent tool in ascertaining and promoting what a well-trained clinical pharmacist can contribute to the health care through patient centered practice. Currently, there are a great number of clinical pharmacists who are wasting their knowledge and skill in a routine and traditional way of dispensing despite they are well trained to provide a patient centered care which in turn curb many limitations of a traditional way of dispensing with a minimal patient contact time and provision of in adequate information to them.

Despite the importance of clinical pharmacists services to the improvement of asthma outcomes, clinical pharmacists face many challenges in the involvement of asthma patients, such as poor awareness among general public, lack of specific legislation and recognition from other health care providers Previously done studies have shown that clinical pharmacist led interventions had improvements in asthma outcomes. However, evidence for different interventions is not totally conclusive; Therefore, the present randomized controlled trial will set up to study the hypothesis that such pharmacist intervention will result in an improved asthma control in adult patients over a 6-month period.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Physician's diagnosis of asthma

Exclusion Criteria:

* Participation in another asthma education program
* Pregnancy
* Communication difficulties
* Seasonal asthma (asthma symptoms that only occur in a seasonal pattern)
* Other pathologies such as COPD, emphysema, lung cancer, respiratory infection
* Terminal illness (any disease that is reasonably expected to result in the patient's death)
* Having an asthma control test level of <15 (indicating seriously uncontrolled asthma; for ethical reasons, these patients will be immediately referred ) or
* Having an asthma control test level equaling 25 (indicating complete asthma control; no room for improvement) will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Change in the level of asthma control | change in asthma control at 1,3 and 6 month
  A blinded investigator will assess change in asthma control using the Asthma control test score (ACT). This is a clinically validated asthma control measure that consists of five questions with five alternative responses (classified by decreasing level of asthma control, scored from 5 to 1). The ACT score (range 5-25) is calculated by adding the responses to the five questions; the higher the score, the better asthma control. The ACT will be completed at randomization, as well as 1, 3, and 6 months later. Patients with a maximum score of 25 will be considered "completely controlled," while those with an ACT score of 20-24 will be considered as having "well-managed" asthma, and those with a score of 15-19 will be categorized as "uncontrolled" asthma.

SECONDARY OUTCOMES:
Number of exacerbations of asthma | 6 month
  Asthma exacerbation is one that necessitates the use of oral glucocorticoids, as well as a trip to the emergency room or hospitalization
Improvement in Adherence level | 6 month
  Two validated measures of adherence will be used to assess adherence throughout the study: prescription refill rates and self reporting. During the trial period, the number of units of controller medicine provided to each patient will be documented, and adherence will be computed. The test of adherence to inhaler instrument (TAI) will be used to assess self reported adherence at the end of the trial (TAI).) The TAI is a reliable and homogeneous questionnaire to identify easily non-adherence and to classify from a clinical perspective the barriers related to the use of inhalers in asthma TAI scores 50, 46-49 and less than 45 will be considered as adherent, intermediate adherent and non-adherent respectively.
Change in Inhalation technique skill | 6 month
  The inhalation technique will be rated using an eight-point checklist for metered dosage inhalers (MDI). One point will be awarded for each correct step, and the total score for the inhalation technique will be given as a percentage of correct steps. Patients who make serious inhalation technique errors (failure to remove cap and/or shake MDI; failure to load device and/or inhale fast and deeply via device ) will be given a sum score of zero. For ethical reasons, such major errors will also be corrected in patients belonging to the control group. Good MDIs use technique: when patients respond to greater than or equal to seven the mean score of MDIs use technique (≥70%). Poor MDIs use technique: when patients respond to less than seven the mean score of MDIs use technique (< 70%).
change in Knowledge about disease and treatment | 6 month
  An updated version of the Knowledge of Asthma and Asthma Medicine questionnaire will be used to assess patients' knowledge of asthma and its treatment at the start of the intervention period and after the 6-month follow-up.
Number of Drug therapy problems reduced | 6 month
  Using the PCNE(Pharmaceutical Care Network Europe) Classification tool Version 6.2 from Pharmaceutical Care Network Europe (PCNE) drug therapy problems will be identified. The PCNE V 6.2 has four primary issue domains, eight primary cause domains, and five primary intervention domains. There are 37 grouped sub-domains for causes, 9 grouped sub-domains for problems, and 17 grouped sub-domains for effects.Pharmaceutical care evaluation will be carried out and any drug therapy problems will be addressed accordingly.
Change in Asthma Quality of life | 6 month
  Asthma-specific quality of life will be assessed at the start of the intervention period and after the 6-month follow-up period using the Standardized Asthma Quality of Life Questionnaire (AQLQ(S)).

CONTACTS AND LOCATIONS:
Overall Officials: Eden A Mehari, Msc, Principal Investigator — University of Gondar
Locations (1):
- University of Gondar Specialized and Comprehensive Hospital, Gonder, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
A deidentified analytical dataset will be posted in an open access repository upon study completion.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The time frame will start from the time when summary data are published or start 6 months after publication.
Access Criteria: PD and additional supporting data information will be shared through open-access journals.